CLINICAL TRIAL: NCT01263821
Title: Image Guided Adaptive Multi-modality Therapy in the Treatment of Gliomas
Brief Title: Image Guided Therapy in the Treatment of Gliomas
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 09-0069
Record Dates: First submitted 2010-12-16; First posted 2010-12-21 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Glioma
Keywords: glioma; biologic imaging; magnetic resonance spectroscopy; magnetic resonance imaging; perfusion imaging; diffusion imaging; functional magnetic resonance imaging; radiation therapy; intensity modulated radiation therapy
MeSH Terms: conditions — Glioma | interventions — Magnetic Resonance Spectroscopy; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm I (Experimental): Patients undergo magnetic resonance spectroscopic imaging, functional magnetic resonance imaging (MRI), diffusion-weighted MRI, and perfusion-weighted MRI. Patients then undergo maximum surgical resection followed by intensity-modulated radiation therapy (IMRT) 5 days a week for 6 weeks.
  Interventions: Procedure: Diffusion-weighted magnetic resonance imaging; Procedure: Perfusion-weighted magnetic resonance imaging; Procedure: Functional magnetic resonance imaging; Procedure: Magnetic resonance spectroscopic imaging; Procedure: Therapeutic conventional surgery; Procedure: Quality-of-life assessment; Procedure: Radiation therapy treatment planning/simulation; Procedure: Intensity-modulated radiation therapy; Other: Questionnaire administration

INTERVENTIONS:
Procedure: Diffusion-weighted magnetic resonance imaging — Undergo diffusion-weighted MRI
  Other Names: Diffusion-weighted MRI
Procedure: Perfusion-weighted magnetic resonance imaging — Undergo perfusion-weighted magnetic resonance imaging
  Other Names: Perfusion-weighted MRI
Procedure: Functional magnetic resonance imaging — Undergo functional MRI
  Other Names: fMRI, functional MRI
Procedure: Magnetic resonance spectroscopic imaging — Undergo MR spectroscopic imaging
  Other Names: 1H-nuclear MRSI, Proton MRSI
Procedure: Therapeutic conventional surgery — Undergo maximal surgical resection
Procedure: Quality-of-life assessment — Ancillary studies
Procedure: Radiation therapy treatment planning/simulation — Undergo IMRT planning
Procedure: Intensity-modulated radiation therapy — Undergo intensity-modulated radiation therapy
  Other Names: IMRT
Other: Questionnaire administration — Ancillary studies

SUMMARY:
RATIONALE: New imaging techniques using magnetic resonance imaging give better tumor definition, thus may lead to better tumor targeting and avoid damaging critical parts of normal brain.

PURPOSE: This phase I/II trial is studying how well image-guided therapy works in treating patients with newly diagnosed intracranial glioma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To correlate the imaging findings with pathological grade following surgery in patients with newly diagnosed intra-cranial gliomas.

SECONDARY OBJECTIVES:

I. To determine the feasibility of defining the optimal target volume for radiation therapy using MR spectroscopy, diffusion, perfusion and functional imaging. II. To monitor therapeutic responses following treatment using MR spectroscopy, diffusion imaging and perfusion study.

III. To monitor changes in neurocognitive functioning following image guided therapy.

OUTLINE: Patients undergo magnetic resonance spectroscopic imaging, functional magnetic resonance imaging (MRI), diffusion-weighted MRI, and perfusion-weighted MRI. Patients then undergo maximum surgical resection followed by intensity-modulated radiation therapy (IMRT) 5 days a week for 6 weeks. After completion of study treatment, patients are followed up every 3 months for the first year then every 6 months for another year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, newly diagnosed intracranial glioma
* A diagnostic contrast enhanced CT/MRI demonstrating the lesion prior to registration
* Karnofsky performance status >= 60
* Ability to undergo MR imaging with the use of Gadolinium dye
* Patient must sign a study specific informed consent form; if the patient's mental status precludes his/her giving informed consent, written informed consent may be given by the patient's legal representative

Exclusion Criteria:

* Inability to obtain histological proof of glioma
* Allergy to Gadolinium contrast
* Any condition including metallic implants or cardiac pace makers that make the candidate ineligible for MR imaging
* Any medical condition including renal or cardiac insufficiency that make the candidate a high risk for gadolinium contrast administration
* Karnofsky performance status of =< 50
* Prior history of radiation therapy to the brain
* Pregnancy

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Feasibility of identifying low grade and high grade tumor location with imaging techniques that include MRSI,perfusion MRI, and DTI | Twice a year, after enrollment of first 25 patients, and at study completion

SECONDARY OUTCOMES:
Incorporate imaging techniques of MRSI, perfusion MRI and DTI into the radiotherapy treatment planning system for target delineation | Twice a year, after enrollment of first 25 patients, and at study completion
Clinical efficacy of this biological image-guided treatment in gliomas | Twice a year, after enrollment of first 25 patients, and at study completion

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Silverman, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Cancer Institute, New York, New York, United States